CLINICAL TRIAL: NCT04175353
Title: Tailored Food Solutions for Improving Nutrition and Well-being in Older People: Effects on Postprandial Responses
Brief Title: Effects of Dairy- and Berry-based Snacks on Postprandial Glucose Metabolism in Older People
Acronym: MAVIRE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MAVIRE2 247124; 4249/31/2014 (Other Grant/Funding Number: Tekes)
Record Dates: First submitted 2019-11-14; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Postprandial Hyperglycemia
Keywords: older people; nutrition; dairy; berries; postprandial; glucose; insulin
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dairy snack (Experimental): Drink high in milk protein, 250 ml
  Interventions: Dietary Supplement: Dairy snack
- Orange juice (Active Comparator): Regular orange juice, 250 ml
  Interventions: Dietary Supplement: Dairy snack
- Berry snack 1 (Experimental): Bilberry-blackcurrant purée, 139 g
  Interventions: Dietary Supplement: Berry snack
- Berry snack 2 (Experimental): Lingonberry purée, 122 g
  Interventions: Dietary Supplement: Berry snack
- Berry soup (Active Comparator): Bilberry soup, 250 ml
  Interventions: Dietary Supplement: Berry snack

INTERVENTIONS:
Dietary Supplement: Dairy snack — The effects of dairy snack are compared with orange juice.
  Arms: Dairy snack; Orange juice
Dietary Supplement: Berry snack — The effects of two berry snacks are compared with berry soup.
  Arms: Berry snack 1; Berry snack 2; Berry soup

SUMMARY:
Malnutrition or its risk is common among older people. To maintain adequate nutrition, increased meal frequency is important. In addition to main meals, regular consumption of nutrient- and energy-dense snacks is recommended. The study examines the post-meal responses to dairy- and berry-based snacks tailored for older people. The plasma concentrations of glucose, insulin and free fatty acids are measured during three hours after snack consumption. In addition, subjective satiety responses and heart rate variability are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Home-dwelling

Exclusion Criteria:

* Smoking
* Type 1 diabetes
* Type 2 diabetes treated with oral medications or insulin
* Cognitive impairment
* Antibiotic medication within the past 3 months
* Blood donation within the past month

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in postprandial glucose | 3 hrs
  Changes in plasma glucose concentration within 3 hrs after meal
Change in postprandial insulin | 3 hrs
  Changes in plasma insulin concentration within 3 hrs after meal

SECONDARY OUTCOMES:
Change in postprandial free fatty acids | 3 hrs
  Changes in plasma free fatty acid concentration within 3 hrs after meal
Change in postprandial satiety scores assessed by using visual analogy scales | 3 hrs
  Visual analogue scales (VAS) are used to assess satiety and other related subjective sensations (fullness, hunger, desire to eat, alertness) within 3 hrs after meal. Each VAS consists of a 100-mm horizontal line anchored with verbal descriptions at each end expressing the weakest (0 mm) or strongest (100 mm) statement of sensation. Results are scores between 0 and 100.
Heart rate variability | 3 hrs
  Electrocardiography monitoring for assessment of several variables of heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Törrönen, PhD, Principal Investigator — University of Eastern Finland, Institute of Public Health and Clinical Nutrition; Marjukka Kolehmainen, Professor, Principal Investigator — University of Eastern Finland, Institute of Public Health and Clinical Nutrition; Mika Tarvainen, PhD, Principal Investigator — University of Eastern Finland, Department of Applied Physics
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torronen R, Jarvinen S, Kolehmainen M. Postprandial glycemic responses to a high-protein dairy snack and energy-enriched berry snacks in older adults. Clin Nutr ESPEN. 2022 Oct;51:231-238. doi: 10.1016/j.clnesp.2022.08.026. Epub 2022 Aug 30. PMID 36184209